CLINICAL TRIAL: NCT06766474
Title: Bupivacaine Hydrochloride-Soaked Dressing Versus Subcutaneous Infiltration for Postoperative Analgesia in Skin Graft Donor Site: a Randomized Controlled Clinical Trial
Brief Title: The Rule of Bupivacaine Hydrochloride in Skin Graft Donor Site
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, MOHAMED SABRY, lecturer of plastic and reconstructive surgery, Minia University, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bupivacaine analgesia
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Skin Graft Complications; Pain Management
Keywords: bupivacaine; skin graft; pain; donor site; local anesthesia
MeSH Terms: conditions — Agnosia; Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group I (soaked dressing group) (Experimental): the donor site dressing was kept soaked in an aqueous solution of bupivacaine HCL in a concentration of 0.25%.
  Interventions: Drug: Bupivacain
- Group II (subcutaneous infiltration group) (Experimental): Subcutaneous infiltration of the study medication.
  Interventions: Drug: Bupivacain
- Group III (control group) (No Intervention): the conventional dressing was applied without any adjectives

INTERVENTIONS:
Drug: Bupivacain — to our knowledge, this study is the 1st to compare the efficacy of bupivacaine hydrochloride-soaked dressing versus subcutaneous infiltration for postoperative donor site pain control for patients undergoing STSG procedures.
  Arms: Group I (soaked dressing group); Group II (subcutaneous infiltration group)

SUMMARY:
Split Thickness Skin Graft is frequently utilized for reconstructing skin loss of various causes. Unfortunately, the donor site of the STSG has an unavoidable, annoying post-operative pain

DETAILED DESCRIPTION:
The primary objective of this study was to compare the efficacy of bupivacaine hydrochloride-soaked dressing versus bupivacaine HCL subcutaneous infiltration for postoperative donor site pain control for patients undergoing STSG procedures. The patients were divided in 3 equal groups, investigated soaked dressing vs subcutaneous infiltration vs conventional dressing .

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status classification I-II
* scheduled for STSG harvested from a single thigh donor site to reconstruct skin loss post burn or trauma

Exclusion Criteria:

* uncooperative
* refusing patient,
* under immunosuppressive treatment
* diabetics
* lower-limb neuropathy
* under corticosteroids treatment
* allergy to the study drug,
* STSG procedures performed under spinal anesthesia
* pregnancy
* had a history of opioid abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
screening pain | 24 hours
  Numerical rating scale (NRS), 0, 1, 2, 4, 8, 12, 18 and 24h, a tool for screening pain, often utilized to evaluate pain intensity on a 0-10 scale, where zero indicates no pain and 10 signifies the worst pain possible, in the 1st 24h postoperatively
frequency of analgesia and the fentanyl requirement | 24 hours
  1g of paracetamol IV was given to all patients every 8 h and if NRS >3 in the donor site patient received 30 mg IV of ketorolac (the frequency of analgesia), if the pain still, the patient was given fentanyl 50 mcg per time (fentanyl requirement) in the three studied groups Registration of the frequency of time of 1st analgesia, frequency of analgesia (ketorolac) and the fentanyl requirement over 1st 24 h as (0, 1, 2, 4, 8, 12, 18 and 24h).

SECONDARY OUTCOMES:
side effects | 24 hours
  recording any side effects such as convulsions and myocardial depression.

CONTACTS AND LOCATIONS:
Overall Officials: MOHAMED SABRY, MD, Principal Investigator — Lecturer of plastic and reconstructive surgery; Shadwa Rabea, MD, Principal Investigator — Assistant professor of anesthesia and Intensive Care; Mohab Elsayed, Phd, Principal Investigator — Assistant lecturer of plastic and reconstructive surgery
Locations (1):
- Minia University Hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shahzad F. Management of skin graft donor site in pediatric patients with tumescent technique and AQUACEL(R) Ag foam dressing. J Plast Surg Hand Surg. 2021 Oct;55(5):309-314. doi: 10.1080/2000656X.2021.1883632. Epub 2021 Feb 16. PMID 33591240
- [Background] Liu SS, Richman JM, Thirlby RC, Wu CL. Efficacy of continuous wound catheters delivering local anesthetic for postoperative analgesia: a quantitative and qualitative systematic review of randomized controlled trials. J Am Coll Surg. 2006 Dec;203(6):914-32. doi: 10.1016/j.jamcollsurg.2006.08.007. Epub 2006 Oct 25. No abstract available. PMID 17116561
- [Background] Sinha S, Schreiner AJ, Biernaskie J, Nickerson D, Gabriel VA. Treating pain on skin graft donor sites: Review and clinical recommendations. J Trauma Acute Care Surg. 2017 Nov;83(5):954-964. doi: 10.1097/TA.0000000000001615. PMID 28598907
- [Background] Bittner EA, Shank E, Woodson L, Martyn JA. Acute and perioperative care of the burn-injured patient. Anesthesiology. 2015 Feb;122(2):448-64. doi: 10.1097/ALN.0000000000000559. PMID 25485468
- [Background] Akan M, Yildirim S, Misirlioglu A, Ulusoy G, Akoz T, Avci G. An alternative method to minimize pain in the split-thickness skin graft donor site. Plast Reconstr Surg. 2003 Jun;111(7):2243-9. doi: 10.1097/01.PRS.0000060087.93322.2F. PMID 12794466